CLINICAL TRIAL: NCT04892498
Title: A Prospective Multicenter Clinical Study of Hypofractionated Radiotherapy Combined With PD-1 Inhibitor Sequential GM-CSF and IL-2 for the Treatment of Advanced Refractory Solid Tumors
Brief Title: Hypofractionated Radiotherapy Combined With PD-1 Inhibitor Sequential GM-CSF and IL-2 for the Treatment of Advanced Refractory Solid Tumors (PRaG2.0)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JD-LK-2021-035-01
Record Dates: First submitted 2021-04-19; First posted 2021-05-19 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2021-08

CONDITIONS: Advanced Refractory Solid Tumors
Keywords: hypofractionated radiotherapy; PD-1 inhibitor; GM-CSF; IL-2
MeSH Terms: interventions — Radiation Dose Hypofractionation; Immune Checkpoint Inhibitors; Granulocyte-Macrophage Colony-Stimulating Factor; Interleukin-2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RT+PD-1+GM-CSF+IL-2 (Experimental)
  Interventions: Radiation: Hypofractionated radiotherapy; Drug: PD-1 inhibitor; Drug: GM-CSF; Drug: IL-2

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — 10-24Gy/5-8Gy/2-3f
Drug: PD-1 inhibitor — q3w, until PD
Drug: GM-CSF — 200μg, D1-D7, ≥8 cycles
Drug: IL-2 — at a dose of 2 million IU, D8-D14, ≥8 cycles

SUMMARY:
This is a prospective multicenter clinical study to determine the efficacy and safety of hypofractionated radiotherapy combined with PD-1 inhibitor sequential GM-CSF and IL-2 for advanced multiple metastatic solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. The enrolled patients meet the recurrence or metastasis of advanced solid malignant tumors, have a clear pathological diagnosis report or medical history, the guidelines do not clearly recommend standard treatment plans or cannot tolerate standard treatment plans, and have clear measurable metastatic lesions (>1cm);
3. No congestive heart failure, unstable angina, or unstable arrhythmia occurred in the past 6 months.
4. The patient's activity status score is 0-3 points based on the Eastern Cooperative Oncology Group (ECOG) scoring method, and the life expectancy assessment is ≥3 months.
5. No serious hematopoietic function, abnormal heart, lung, liver, kidney function and immune deficiency in the past.
6. One week before admission, the absolute value of T lymphocytes was ≥0.5 times the lower limit of normal, and neutrophils ≥1.0×109/L; AST and ALT were ≤3.0 times the upper limit of normal (for liver cancer/liver metastasis ≤5.0 times) Upper limit of normal); creatinine ≤3.0 times the upper limit of normal.
7. The patient have the ability to understand and voluntarily sign an informed consent form.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Those with a history of other malignant diseases in the last 5 years, except for cured skin cancer and cervical carcinoma in situ.
3. If there is a history of uncontrolled epilepsy, central nervous system disease or mental disorder, the investigator's judgment of its clinical severity may hinder the signing of informed consent or affect the patient's compliance with medication.
4. Clinically serious (ie active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) grade II or more severe congestive heart failure, or severe arrhythmia requiring drug intervention, or recent A history of myocardial infarction within 12 months.
5. Those who need immunosuppressive therapy for organ transplantation.
6. A known major active infection, or the researcher's judgment has major blood, kidney, metabolism, gastrointestinal, endocrine function or metabolic disorders, or other serious uncontrolled accompanying diseases.
7. Those who are allergic to any research drug ingredients.
8. A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation, or those with other immune-related diseases that require long-term oral hormone therapy.
9. In the period of acute and chronic tuberculosis infection (T-spot test is positive, patients with suspected tuberculosis foci on chest X-ray).
10. Other situations that the researcher thinks are not suitable for inclusion in the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-05-30 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
progression free survival，PFS | Up to 3 years
  Time from cycle 1, day 1 of treatment to disease progression or death due to any cause

SECONDARY OUTCOMES:
Overall response rate，ORR | Up to 3 years
  The proportion of patients with at least one tumor scan of complete response (CR) or partial response (PR) using RECIST v1.1.
Disease control rate，DCR | Up to 3 years
  The proportion of patients with at least one tumor scan of complete response (CR) or partial response (PR) or stable disease (SD) using RECIST v1.1.
Overall survival，OS | Up to 3 years
  Time from cycle 1, day 1 of treatment until death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Liyuan Zhang, Dr, Principal Investigator — Second Affiliated Hospital of Soochow University
Locations (16):
- China (16):
  - Peking University Third Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - Xiangya Hospital of Central South University, Changsha
  - Chongqing University Cancer Hospital, Chongqing
  - The Sixth Affiliated Hospital ，Sun Yat-seen University, Guangzhou
  - Cancer Hospital of The University of Chinese Academy of Sciences, Hangzhou
  - The First Affiliated Hospital of USTC, Hefei
  - Shandong Provincial Tumor Hospital, Jinan
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Cancer Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Second Affiliated Hospital of Soochow University, Suzhou
  - Renmin Hospital of Wuhan University, Wuhan
  - Jiangyin People's Hospital, Wuxi
  - The Affilated Hospital of Xuzhou Medical University, Xuzhou